CLINICAL TRIAL: NCT02274233
Title: Multicenter, Open-label, Dose-escalation Study of SP-420 in Subjects With Transfusion-dependent β-Thalassemia
Brief Title: Safety and Pharmacokinetic Study of Escalating Doses of SP-420, an Iron Chelator, in Patients With β-Thalassemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Changes in renal function parameters.
Sponsor: Sideris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-420-702
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Iron Overload; Beta-Thalassemia
Keywords: Chelation; Iron Overload; Thalassemia; Transfusion; Iron Chelation
MeSH Terms: conditions — Iron Overload; beta-Thalassemia; Thalassemia | interventions — SP-420

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1.5 mg/kg (Experimental): 1.5 mg/kg SP-420 once daily for 14 days
  Interventions: Drug: SP-420
- 3 mg/kg (Experimental): 3 mg/kg SP-420 once daily for 14 days
  Interventions: Drug: SP-420
- 6 mg/kg (Experimental): 6 mg/kg SP-420 once daily for 14 days
  Interventions: Drug: SP-420
- 12 mg/kg (Experimental): 12 mg/kg SP-420 once daily for 14 days
  Interventions: Drug: SP-420
- 24 mg/kg (Experimental): 24 mg/kg SP-420 once daily for 28 days
  Interventions: Drug: SP-420
- 9 mg/kg (Experimental): 9 mg/kg SP-420 twice daily for 28 days
  Interventions: Drug: SP-420

INTERVENTIONS:
Drug: SP-420

SUMMARY:
The purpose of this study is to assess safety and amount of the study drug in the blood after increasing doses of SP-420. The study will be conducted in patients with β-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has iron-overload secondary to β-thalassemia requiring chronic red blood cell transfusions and iron chelation therapy
* Subject weighs ≥35 kg
* Subject is willing to discontinue current iron chelation therapy at least 7 days prior to the first dose of SP-420 and for the duration of the study
* Serum ferritin ≥700 ng/mL and iron saturation ≥70% within 3 weeks before Baseline (Day 1)
* Cardiac T2* score >20 msec within 6 months before Baseline (Day 1)
* Willing to use contraception during the study

Exclusion Criteria:

* Pregnant or breast-feeding
* Serum creatinine greater than the upper limit of normal
* Platelet count <100 × 10^9/L
* Use of another investigational drug within the last 30 days
* Significant cardiac, renal, hepatic dysfunction or other clinically significant conditions that, in the opinion of the Investigator, would exclude the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 35 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SP-420 | Day 7
Area under the plasma concentration versus time curve (AUC) of SP-420 | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Sideris Pharmaceuticals, Inc. Sideris Pharmaceuticals, Inc., Study Director — Sideris Pharmaceuticals, Inc.
Locations (7):
- United States (3):
  - Sideris Investigative Site, Boston, Massachusetts
  - Sideris Investigative Site, New York, New York
  - Sideris Investigative Site, Philadelphia, Pennsylvania
- Sideris Investigative Site, Toronto, Ontario, Canada
- Sideris Investigative Site, Beirut, Lebanon
- Sideris Investigative Site, Bangkok, Thailand
- Sideris Investigative Site, Izmir, Turkey (Türkiye)